CLINICAL TRIAL: NCT05067829
Title: Comparison of the Effect of Rocuronium Dosing Based on Ideal, Corrected or Total Body Weight on Rapid Sequence Intubation With Priming on Neuromuscular Blockage and Intubation Condition in Elderly Patients.
Brief Title: Rapid Sequence Intubation With Rocuronium in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, aysun postaci, Associate Prof. Dr, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E1-21-1849
Record Dates: First submitted 2021-09-24; First posted 2021-10-05 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Rapid Sequence Induction; Rapid Sequence Intubation; Rocuronium
Keywords: Rapid Sequence Induction and Intubation; Rapid Sequence Intubation; Rocuronium; Geriatrics
MeSH Terms: interventions — Neuromuscular Monitoring

STUDY DESIGN:
Intervention Model Description: Prospective randomized contrrolled study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ideal Body weight (Active Comparator): ROCURONIUM PRIMING DOSE 0,06 MG/KG FOR IDEAL BODY WEIGHT BEFORE 3 MINUTES BEFORE INDUCTION.
  AFTER INDUCTION, ROCURONIUM 0,94 MG/KG FOR IDEAL BODY WEIGHT WILL BE GIVEN.
  Interventions: Device: Train of four(TOF)
- Total Body Weight (Active Comparator): ROCURONIUM PRIMING DOSE 0,06 MG/KG FOR TOTAL BODY WEIGHT BEFORE 3 MINUTES BEFORE INDUCTION.
  AFTER INDUCTION, ROCURONIUM 0,94 MG/KG FOR TOTAL BODY WEIGHT WILL BE GIVEN.
  Interventions: Device: Train of four(TOF)
- Corrected Body Weight (Active Comparator): ROCURONIUM PRIMING DOSE 0,06 MG/KG FOR CORRECTED BODY WEIGHT BEFORE 3 MINUTES BEFORE INDUCTION.
  AFTER INDUCTION, ROCURONIUM 0,94 MG/KG FOR CORRECTED BODY WEIGHT WILL BE GIVEN.
  Interventions: Device: Train of four(TOF)

INTERVENTIONS:
Device: Train of four(TOF) — Train of four(TOF) monitoring after anesthesia induction

SUMMARY:
With the prolongation of life expectancy, the frequency of surgical intervention and anesthesia increases in elderly patients. The rapid Sequence Intubation(RSI) technique is preferred in patients with aspiration risk and who will undergo general anesthesia, especially in the pandemic period, to reduce or eliminate the aerosolization of respiratory secretions. The use of rocuronium at a dose of 1 mg/kg in RSI also causes prolongation of the recovery of neuromuscular block. This study aimed to compare the intubation conditions and train-of-four count(TOFC) 1-2 times of the rocuronium doses with priming according to ideal body weight(IBW), corrected body weight(CBW), and total body weight(TBW) in RSI of patients aged >65 years.

DETAILED DESCRIPTION:
The number of elderly patients (>65 y) increases, and a large proportion of these patients will require surgery and anesthesia at some point. Changes in the neuromuscular junction, organ systems, and cardiac output that occur with aging cause changes in response to neuromuscular blockers. One of the reasons for rapid sequence intubation(RSI) preference is to reduce or eliminate aerosolization of respiratory secretions during general anesthesia and airway manipulation in surgical cases during the pandemic period. Guidelines regarding this subject recommend securing the airway quickly with RSI, and it is reported that aerosol production would decrease with this method. This study aimed to compare the intubation conditions and the train-of-four count (TOFC) 1 and 2 response times of the patients aged 65 and above, who were administered rocuronium at a priming dose (0.06 mg/kg) according to ideal body weight(IBW), corrected body weight(CBW), and total body weight (TBW) before induction, followed by administration of 0.94 mg/kg rocuronium 3 minutes after the anesthesia induction and intubated 45 seconds later.

ELIGIBILITY:
Inclusion Criteria:

* Elective abdominal surgery
* Age > 65 years
* ASA I-II -III

Exclusion Criteria:

* Patient with history of allergy to rocuronium
* Body Mass Index > 35 kg/m2
* Patient who had history of difficult intubation or high possibility of difficult intubation
* Neuromuscular disease
* Kidney failure (GFR < 30 ml/dk/m2)

Ages: 65 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 75 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The percent of excellent intubation condition | During intubation from start to finish of the study
  Score 1: Poor jaw relaxation/ Active resistance to blade/closing vokal kord/ Severe coughing or bucking/ Vigorous limb movement Score 2: Acceptable jaw relaxation/ Intermediate vokal cord moving/ slight limb and diaphram movement score 3: relaxed laryngoscopy/ abducted vocal cords/ no limb and diphragm movement
TOF value during intubation procedure | During intubation from start to finish of the study
  Train of four monitoring during induction and intubation
Time to TOFR equal to zero | During intubation from start to finish of the study
  Time from rocuronium induction to TOFR equal to zero
Time to TOFC equal to 1 | During intubation from start to finish of the study
  Time from rocuronium induction to TOFc equal to 1

CONTACTS AND LOCATIONS:
Overall Officials: Nadide Aysun Postacı, Principal Investigator — aysunposta@yahoo.com
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No